CLINICAL TRIAL: NCT00193063
Title: Phase II Trial of Weekly Gemcitabine and Herceptin in the Treatment of Patients With HER-2 Overexpressing Metastatic Breast Cancer
Brief Title: Weekly Gemcitabine and Trastuzumab in the Treatment of Patients With Human Epidermal Growth Factor Receptor 2 (HER2) Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 44
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients entering this trial received treatment with a combination of gemcitabine and trastuzumab. Gemcitabine 1000 mg/m2 was administered intravenously on days 1, 8,and 15 of a 28-day cycle. Trastuzumab was administered as a 4 mg/kg intravenous loading dose on day 1 and subsequently at a dose of 2 mg/kg on a weekly basis.
  Interventions: Drug: Trastuzumab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab
  Other Names: Herceptin
Drug: Gemcitabine — Gemcitabine
  Other Names: Gemzar

SUMMARY:
Due to its remarkable activity as salvage treatment in women with metastatic breast cancer as well as the additive activity observed for gemcitabine administered in combination with trastuzumab, the clinical activity of the combination of gemcitabine administered with trastuzumab represents an exciting and ideal combination to further evaluate in Her 2 over-expressing metastatic breast cancer patients.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

Gemcitabine + Trastuzumab

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Her-2 positive metastatic breast cancer confirmed by biopsy
* Measurable disease
* Able to perform activities of daily living without considerable
* No previous chemotherapy with gemcitabine
* No more than one prior chemotherapy regimen for metastatic breast cancer
* Adequate bone marrow, liver and renal function
* Normal heart function
* Give written informed consent prior to entering this study.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Received previous treatment with gemcitabine
* History of brain metastases
* Serious underlying medical conditions

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-07; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Yardley DA, Burris HA 3rd, Hanson S, Greco FA, Spigel DR, Barton J, Hainsworth JD. Weekly gemcitabine and trastuzumab in the treatment of patients with HER2-overexpressing metastatic breast cancer. Clin Breast Cancer. 2009 Aug;9(3):178-83. doi: 10.3816/CBC.2009.n.029. PMID 19661042
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/q32122204r774032/fulltext.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine/Trastuzumab: All patients entering this trial received treatment with a combination of gemcitabine and trastuzumab. Gemcitabine 1000 mg/m2 was administered intravenously on days 1, 8,and 15 of a 28-day cycle. Trastuzumab was administered as a 4 mg/kg intravenous loading dose on day 1 and subsequently at a dose of 2 mg/kg on a weekly basis.
Period: Overall Study
Arm/Group | Gemcitabine/Trastuzumab
Started | 41
Completed | 37
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine/Trastuzumab
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine/Trastuzumab
Number analyzed (Participants) | 37
percentage of participants | 30 [17 to 46]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 21 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Trastuzumab
Number analyzed (Participants) | 41
months | 4 [1.9 to 5.3]

3. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Trastuzumab
Number analyzed (Participants) | 41
months | 21 [11.5 to 30.5]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 14/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=41)
Confusion (Psychiatric disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Infection - pneumonia (Infections and infestations) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Infection - port site (Infections and infestations) | 2 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Fever (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Infection - urinary tract (Infections and infestations) | 1 (1)
Death NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=41)
Hemoglobin (Blood and lymphatic system disorders) | 33 (104)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (14)
Constipation (Gastrointestinal disorders) | 10 (17)
Diarrhea (Gastrointestinal disorders) | 9 (23)
Fatigue (General disorders) | 35 (125)
Hypertension (Cardiac disorders) | 7 (14)
Hypotension (Cardiac disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (14)
Nausea (Gastrointestinal disorders) | 28 (56)
Stomatitis (Gastrointestinal disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 16 (22)
Anorexia (Gastrointestinal disorders) | 11 (24)
Rigors/chills (General disorders) | 4 (4)
Fever (General disorders) | 13 (16)
Leukocytes (Blood and lymphatic system disorders) | 26 (74)
Mucositis (Gastrointestinal disorders) | 4 (7)
Neutrophils (Blood and lymphatic system disorders) | 28 (67)
Platelets (Blood and lymphatic system disorders) | 25 (69)
Weight loss (General disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.